CLINICAL TRIAL: NCT04613648
Title: Ultrasonographic Assessment of Painful and Stiff Hemiplegic Shoulder in Subacute Stroke Patients in Terms of Adhesive Capsulitis
Brief Title: Ultrasonographic Assessment of Painful and Stiff Hemiplegic Shoulder in Terms of Adhesive Capsulitis
Status: Terminated | Type: Observational
Why Stopped: The study was stopped because the sample size calculated a priori could not be reached within the study period.
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ilker şengül, Principal Investigator, Izmir Katip Celebi University
Other Study IDs: 2020-GOKAE-0356
Record Dates: First submitted 2020-10-22; First posted 2020-11-03 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Adhesive Capsulitis of the Shoulder; Hemiplegia
Keywords: Shoulder; Hemiplegia; Adhesive capsulitis
MeSH Terms: conditions — Bursitis; Hemiplegia | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Painful and stiff hemiplegic side shoulders of stroke patients
  Interventions: Diagnostic Test: Imaging
- Group B: Asymptomatic non-hemiplegic side shoulders of stroke patients
  Interventions: Diagnostic Test: Imaging
- Group C: Non-dominant side shoulders of healthy volunteers
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — Ultrasonographic imaging of the shoulder

SUMMARY:
Although a relationship has been reported between stroke and adhesive capsulitis, it is controversial whether the underlying cause of the capsular changes seen in hemiplegic shoulder pain is true adhesive capsulitis. Although there has been a limited number of studies, ultrasound, which has been reported as a sensitive and specific method in the diagnosis of true (idiopathic) adhesive capsulitis, has not yielded similar results to arthrography and MRI in demonstrating fibrotic and adhesive changes in the glenohumeral capsule in stroke patients with hemiplegic shoulder pain. This study aims to investigate ultrasonographic structural changes that may be associated with adhesive capsulitis in subacute stroke patients with painful and stiff hemiplegic side shoulder.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain is one of the commonly seen complications of a stroke. Limitation of shoulder joint movement is added to hemiplegic shoulder pain in time. Therefore, adhesive capsulitis is one of the differential diagnoses that come to mind first in patients with hemiplegic shoulder pain and stiffness. Indeed, in arthrographic and magnetic resonance imaging (MRI) studies, it has been reported that adhesive capsulitis (or more accurately, capsular changes), is quite frequent.

Although a relationship has been reported between stroke and adhesive capsulitis, it is controversial whether the underlying cause of the capsular changes seen in hemiplegic shoulder pain is true adhesive capsulitis. Although these capsular changes and joint limitations in patients with hemiplegic shoulder pain may theoretically be related to idiopathic adhesive capsulitis, secondary causes including spasticity, contracture, fibrosis due to lack of movement, rotator cuff lesions, and glenohumeral subluxation have also been emphasized as a cause of the capsular restriction. Although there have been a limited number of studies, ultrasound, which has been reported as a sensitive and specific method in the diagnosis of true (idiopathic) adhesive capsulitis, has not yielded similar results to arthrography and MRI in demonstrating fibrotic and adhesive changes in the glenohumeral capsule in stroke patients with hemiplegic shoulder pain and stiffness. Because ultrasonographic examinations are mostly focused on rotator cuff tendons, bicipital tendon, and subacromial bursa, lack of detailed examination in terms of adhesive capsulitis may be one of the underlying reasons for this inconsistency. In this context, this study aims to investigate ultrasonographic structural changes that may be associated with adhesive capsulitis in subacute stroke patients with painful and stiff hemiplegic side shoulder.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Stroke duration from 1 month to 6 months
* To be able to communicate well
* Presence of hemiplegic side shoulder pain
* Limitation of passive glenohumeral joint abduction on the hemiplegic side
* Limitation of passive glenohumeral joint external rotation of the hemiplegic side

Exclusion Criteria:

* Stroke duration <1 month or > 6 months
* Only presence of one of the pain or stiffness in the hemiplegic side shoulder
* History of pre-stroke shoulder pain independent from the side of shoulder
* Pain and / or stiffness in the non-hemiplegic side shoulder
* History of shoulder injury (independent from the side)
* History of upper extremity surgery (independent from the side)
* Weakness in both upper extremities
* Existence of non-stroke diseases (osteoarthritis, inflammatory arthritis, etc.) that may cause restriction in the shoulder joint
* Inability to communicate properly
* <40 years old
* Hand pain and/or swelling in addition to shoulder pain and stiffness,

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subacute stroke patients with painful and stiff shoulder in the hemiplegic side, and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Coracohumeral ligament thickness | Through study completion, an average of 3 year
  The thickness in mm of the thickest part of the coracohumeral ligament on the axial-oblique plane with the shoulder in the neutral position
Soft tissue composition of the rotator interval | Through study completion, an average of 3 year
  The presence of soft tissue increase (hypoechogenic compared to the biceps tendon and hyperechogenic compared to the joint fluid around the biceps tendon) in the imaging of the rotator interval on the transverse oblique plane
Vascularity in the rotator interval | Through study completion, an average of 3 year
  The presence of increased vascularity in the color Doppler sonographic imaging of the rotator interval on the transverse oblique plane

CONTACTS AND LOCATIONS:
Overall Officials: İlker Şengül, M.D., Principal Investigator — İzmir Katip Çelebi University
Locations (1):
- İlker Şengül, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalichman L, Ratmansky M. Underlying pathology and associated factors of hemiplegic shoulder pain. Am J Phys Med Rehabil. 2011 Sep;90(9):768-80. doi: 10.1097/PHM.0b013e318214e976. PMID 21430513
- [Background] Hakuno A, Sashika H, Ohkawa T, Itoh R. Arthrographic findings in hemiplegic shoulders. Arch Phys Med Rehabil. 1984 Nov;65(11):706-11. PMID 6497618
- [Background] Rizk TE, Christopher RP, Pinals RS, Salazar JE, Higgins C. Arthrographic studies in painful hemiplegic shoulders. Arch Phys Med Rehabil. 1984 May;65(5):254-6. PMID 6712451
- [Background] Lo SF, Chen SY, Lin HC, Jim YF, Meng NH, Kao MJ. Arthrographic and clinical findings in patients with hemiplegic shoulder pain. Arch Phys Med Rehabil. 2003 Dec;84(12):1786-91. doi: 10.1016/s0003-9993(03)00408-8. PMID 14669184
- [Background] Tavora DG, Gama RL, Bomfim RC, Nakayama M, Silva CE. MRI findings in the painful hemiplegic shoulder. Clin Radiol. 2010 Oct;65(10):789-94. doi: 10.1016/j.crad.2010.06.001. Epub 2010 Jul 21. PMID 20797464
- [Background] Wilson RD, Chae J. Hemiplegic Shoulder Pain. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):641-55. doi: 10.1016/j.pmr.2015.06.007. Epub 2015 Sep 9. PMID 26522903
- [Background] Manara JR, Taylor J, Nixon M. Management of shoulder pain after a cerebrovascular accident or traumatic brain injury. J Shoulder Elbow Surg. 2015 May;24(5):823-9. doi: 10.1016/j.jse.2014.12.003. Epub 2015 Feb 3. PMID 25660242
- [Background] Wu H, Tian H, Dong F, Liang W, Song D, Zeng J, Ding Z, Shi Y, Luo H, Xu J. The role of grey-scale ultrasound in the diagnosis of adhesive capsulitis of the shoulder: a systematic review and meta-analysis. Med Ultrason. 2020 Sep 5;22(3):305-312. doi: 10.11152/mu-2430. Epub 2020 Apr 14. PMID 32399538
- [Background] Lee IS, Shin YB, Moon TY, Jeong YJ, Song JW, Kim DH. Sonography of patients with hemiplegic shoulder pain after stroke: correlation with motor recovery stage. AJR Am J Roentgenol. 2009 Feb;192(2):W40-4. doi: 10.2214/AJR.07.3978. PMID 19155379
- [Background] Idowu BM, Ayoola OO, Adetiloye VA, Komolafe MA. Sonographic Evaluation of Structural Changes in Post-Stroke Hemiplegic Shoulders. Pol J Radiol. 2017 Mar 13;82:141-148. doi: 10.12659/PJR.899684. eCollection 2017. PMID 28382186
- [Background] Martinoli C, Bianchi S, Prato N, Pugliese F, Zamorani MP, Valle M, Derchi LE. US of the shoulder: non-rotator cuff disorders. Radiographics. 2003 Mar-Apr;23(2):381-401; quiz 534. doi: 10.1148/rg.232025100. PMID 12640155
- [Background] Sabari JS, Maltzev I, Lubarsky D, Liszkay E, Homel P. Goniometric assessment of shoulder range of motion: comparison of testing in supine and sitting positions. Arch Phys Med Rehabil. 1998 Jun;79(6):647-51. doi: 10.1016/s0003-9993(98)90038-7. PMID 9630143
- [Background] MacDermid JC, Chesworth BM, Patterson S, Roth JH. Intratester and intertester reliability of goniometric measurement of passive lateral shoulder rotation. J Hand Ther. 1999 Jul-Sep;12(3):187-92. doi: 10.1016/s0894-1130(99)80045-3. PMID 10459526
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Brunnstrom S. Motor testing procedures in hemiplegia: based on sequential recovery stages. Phys Ther. 1966 Apr;46(4):357-75. doi: 10.1093/ptj/46.4.357. No abstract available. PMID 5907254
- [Background] Homsi C, Bordalo-Rodrigues M, da Silva JJ, Stump XM. Ultrasound in adhesive capsulitis of the shoulder: is assessment of the coracohumeral ligament a valuable diagnostic tool? Skeletal Radiol. 2006 Sep;35(9):673-8. doi: 10.1007/s00256-006-0136-y. Epub 2006 May 25. PMID 16724200
- [Background] Tamborrini G, Moller I, Bong D, Miguel M, Marx C, Muller AM, Muller-Gerbl M. The Rotator Interval - A Link Between Anatomy and Ultrasound. Ultrasound Int Open. 2017 Jun;3(3):E107-E116. doi: 10.1055/s-0043-110473. Epub 2017 Aug 23. PMID 28845477
- [Background] Lee JC, Sykes C, Saifuddin A, Connell D. Adhesive capsulitis: sonographic changes in the rotator cuff interval with arthroscopic correlation. Skeletal Radiol. 2005 Sep;34(9):522-7. doi: 10.1007/s00256-005-0957-0. Epub 2005 Jul 6. PMID 15999280
- [Background] Adey-Wakeling Z, Arima H, Crotty M, Leyden J, Kleinig T, Anderson CS, Newbury J; SEARCH Study Collaborative. Incidence and associations of hemiplegic shoulder pain poststroke: prospective population-based study. Arch Phys Med Rehabil. 2015 Feb;96(2):241-247.e1. doi: 10.1016/j.apmr.2014.09.007. Epub 2014 Sep 28. PMID 25264111